CLINICAL TRIAL: NCT06744387
Title: Tissue Oxygenation Monitoring of Anterolateral Thigh (ALT) Flaps, Using FORE-SIGHT ELITE Near InfraRed Spectroscopy (NIRS) - A Pilot Study
Brief Title: Anterolateral Tigh (ALT) Flaps Oxygenation Monitoring by NIRS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Vera Saldien, MD, University Hospital, Antwerp
Other Study IDs: EDGE 003917
Record Dates: First submitted 2024-11-27; First posted 2024-12-20 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Reconstructive Flap Surgery; Fasciocutaneous Anterolateral Thigh Flap; Postoperative Monitoring; Flap Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with reconstructive flap surgery on upper or lower limb using a fasciocutanous tigh flap
  Interventions: Diagnostic Test: clinical assessments and tissue oxygenation monitoring by Near Infrared Spectroscopy

INTERVENTIONS:
Diagnostic Test: clinical assessments and tissue oxygenation monitoring by Near Infrared Spectroscopy — Flap failure will be identified, based upon gold standard monitoring (flaps skin color, temperature, tissue turgor and capillary refill time) along with Doppler technique during a postoperative period of five days. In all patients Near Infrared Spectroscopy (NIRS) by FORE-SIGHT ELITE will be applied to obtain continuous tissue oxygenation measurements. NIRS values and trends from patients with flap failure (case group) will be compared to NIRS values and trends from patients with no flap failure(control group).

SUMMARY:
The goal of this observational study is to conduct postoperative monitoring in patients who have undergone upper or lower limb reconstructive surgery with an anterolateral thigh flap, by employing the gold standard approach: intermittent assessment of clinical parameters (flap's color, temperature, skin turgor and capillary refill time) combined with Doppler techniques, alongside continuous tissue oxygenation measurements obtained using the CASMED FORE-SIGHT ELITE monitor.The main objective of the study is to provide preliminary data on potential cut-off values indicative of flap failure.

DETAILED DESCRIPTION:
Microvascular reconstructive free flap surgery is commonly used practice in contemporary medicine for managing extensive and complex tissue defects. A primary concern associated with this surgical approach is the risk of flap failure during the postoperative phase, usually resulting from vascular compromise in the first 1-3 days after surgery. Minimizing the time interval to revision surgery enhances the likelihood of salvaging the flap. Hence, effective, and vigilant monitoring is crucial in detecting this feared complication. Currently, the gold standard for monitoring entails the assessment of the flap's skin color, temperature, tissue turgor and capillary refill time, usually supplemented by Doppler techniques. This method of monitoring is labor-intensive and reliant on the expertise of the nursing staff, resulting in variability and inconsistencies. There is a definite need for a more objective, real-time monitoring approach, which is attainable through techniques like Near Infrared Spectroscopy (NIRS). NIRS is a non-invasive tool employed in medical settings to assess regional tissue oxygenation through the placement of specific electrodes at the anatomical site of interest. These electrodes emit photons at multiple wavelengths within the near-infrared spectrum (700-1100 nanometer ) into the tissues and subsequently measure the reflected light patterns. Optical properties of biological molecules alter upon oxygen binding, which causes variations in the near-infrared light absorption patterns. Therefore, the absorption pattern is contingent upon the ratio of oxygenated to deoxygenated hemoglobin. Through analysis of these light patterns and the oxygenated-to-deoxygenated hemoglobin ratio, the NIRS monitor calculates and displays a real-time measurement of tissue oxygen saturation (StO2). This number represents the balance between oxygen supply and uptake in the surrounding tissues and offers information on the underlying hemodynamics. With regards to monitoring after reconstructive flap surgery, NIRS currently occupies a limited role and cannot yet replace the established gold standard of clinical assessment and Doppler techniques. This limited use stems primarily from a lack of consensus on the interpretation of the measured values and the question remains which cut-off values or trends should lead to reintervention. Most of the studies did suggest certain cut-off values, nonetheless, a consensus could not be deduced, except for the ViOptix Tissue Oximeter (ViOptix Inc., Fremont, Ca, USA). An StO2 drop rate of more than 20% per hour during more than 30 minutes could be suggestive of vascular crisis when using this device. Overall, authors attributed the discrepancies in published cut-off values to a lack of large randomized clinical trials and to manufacturer-related variations in the devices, such as number of emitted wavelengths, measuring depth and accuracy, analyzing algorithms.

In this pilot study, we aim to conduct postoperative monitoring in patients who have undergone upper or lower limb reconstructive surgery with an anterolateral thigh flap, employing the gold standard approach for flap surgery, combined with Doppler techniques. Alongside continuous tissue oxygenation measurements will be applied using the FORE-SIGHT ELITE tissue oximeter (FORE-SIGHT ELITE, CAS Medical Systems, Branford, CT USA). The measurements by the FORE-SIGHT ELITE however, remain blinded for the patient and the nursing staff. The data are stored in the FORE-SIGHT ELITE device and will be retrieved after the monitoring period of five days by the investigators. The gold standard approach is used to identify cases of flap failure and distinguish them from control subjects. The 'control' group includes patients with successful flap outcomes and reassuring clinical assessments, while the 'case' group consists of patients with abnormal clinical findings and accompanying flap failure.

The anesthetic management during the reconstructive flap surgery will comply with the standard of care. Each patient will be routinely monitored through pulse oximetry, blood pressure measurements and 5-lead electrocardiography. Patients will be put under general anesthesia using sufentanyl or fentanyl combined with a target-controlled infusion (TCI) of propofol. Muscle paralysis will be induced using rocuronium. Depending on the extensiveness of the operation, a second peripheral line and/or an arterial line for invasive blood pressure measurement and arterial blood gas analysis may be placed. Adequate hemodynamic management is crucial in guaranteeing sufficient perfusion of the flap. Inotropes or vasoactive medications may be employed for this purpose. Body temperature will be monitored and normothermia will be maintained. Following preoperative marking of the flap at the anterolateral thigh (donor site) and identification of dominant vascular branches using Doppler ultrasound, the surgical intervention will be performed. At end of surgery the surgeon marks the location of the main vascular anastomosis sites on the flap for postoperative monitoring of Doppler signals. Two sensors, one at the flap site and one at the donor site, will be attached by the surgeon before departure from the operating room to the Post Anesthetic Care Unit (PACU). Depending on the size of the flap, pediatric sensors will be used. After surgery the patient will stay in the PACU for one night. Continuous NIRS tissue oxygenation measurements will commence upon the patient's arrival at the PACU. The first measurement at the PACU will be considered the baseline value. Trained nurses will conduct hourly clinical assessments of skin color, capillary refill, temperature, skin turgor, and Doppler signals for the first 24 hours. In addition, patients will be routinely monitored with pulse oximetry, 3-lead electrocardiography, and blood pressure measurements. Following their stay in the PACU, patients will be transferred to a regular nursing ward, where the clinical assessment of the flap and the patient's vitals signs monitoring will be continued. In the event of an abnormal clinical evaluation, the nurses will promptly notify the surgeon.

Cases of flap failure will be identified by use of the gold standard(skin color, temperature, tissue turgor and capillary refill time measured by Doppler techniques) along with evaluation of clinical assessments of vital signs while NIRS measurements remain blinded. Following the monitoring period of five days, the stored NIRS values and trends in the FORE-SIGHT ELITE device from both groups will undergo analysis and will be compared. The objective is to gain insight into potential cut-off values for detecting vascular compromise.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for reconstructive flap surgery on either upper or lower limb using a fasciocutaneous anterolateral thigh flap

Exclusion Criteria:

* refusal to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: scheduled for reconstructive flap surgery on either upper or lower limb using a fasciocutaneous anterolateral thigh flap
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
provide preliminary data on potential cut-off values for tissue oxygenation indicative for flap failure | from end of surgery untill five days after surgery
  a decrease of x percent in tissue oxygenation below the baseline value (first measurement upon arrival at the PACU) of the anterolateral thigh flap.
provide preliminary data on potential cut-off values for tissue oxygenation indicative for flap failure | from end of surgery untill five days after surgery
  a decrease of x percent in tissue oxygenation in the anterolateral thigh flap compared to the reference measurements obtained from the unaffected remaining anterolateral thigh.

SECONDARY OUTCOMES:
retrospective time-to-event analysis in patients with flap failure | through study completion, an average of 1 year
  a retrospective time-to-event analysis for the index test (NIRS measurements) and the reference test (the gold standard) within the subgroup of cases with flap failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No